CLINICAL TRIAL: NCT01318720
Title: Short-Term Combined Effects of Thoracic Spine Thrust Manipulation and Cervical Spine Non-Thrust Manipulation in Patients With Mechanical Neck Pain: A RCT
Brief Title: Short-Term Effects of Combined Manual Therapy to the Cervical and Thoracic Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masefield and Cavallaro Physical Therapy (Other)
Responsible Party: Principal Investigator, Michael Masaracchio PT, DPT, PhD(c), OCS, SCS, Senior Staff Physical Therapist, Masefield and Cavallaro Physical Therapy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCPT1
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Neck Pain
Keywords: Neck Pain; Thrust Manipulation; Non-Thrust Manipulation
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Manipulation (Experimental): The experimental group is receiving thoracic spine thrust manipulation and cervical spine non-thrust manipulation.
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Other: Manual Therapy — Thrust manipulation is a type of manual therapy that clinicians apply using a high-velocity, low-amplitude thrust directed at a joint(s)

SUMMARY:
Neck pain continues to be a prevalent condition in our society. Manual therapy (hands on techniques for the treatment of neck pain is an intervention commonly implemented in clinical practice. Recently researchers and clinicians have implemented manual therapy techniques to the thoracic spine (midback) to treat patients with neck pain. To date no studies have examined the short-term combined effects of thoracic spine manual therapy and cervical spine manual therapy in the treatment of patients with mechanical neck pain. The purpose this study is to assess the combined effects of thoracic spine thrust manipulation with cervical spine non-thrust manipulation in patients with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain of less than 3 months
* No symptoms below the shoulder
* Baseline Neck Disability Index score of 10 or greater

Exclusion Criteria:

* Red flags noted in the patient's Medical Screening Questionnaire (i.e. tumor, fracture, metabolic disease, rheumatoid arthritis, osteoporosis, prolonged use of steroid, etc)
* History of whiplash injury within the past two months
* Diagnosis of cervical spinal stenosis
* Uni-lateral or bi-lateral upper extremity radicular symptoms
* Evidence of central nervous system involvement
* Two or more positive neurological signs consistent with nerve root involvement: myotomal muscle weakness, dermatomal sensory loss, diminished or absent reflexes
* Prior surgery to the neck or thoracic spine
* Pending legal action regarding their neck pain, or patients with no fault or workers compensation claims
* Insufficient English language skills to complete the questionnaires
* Inability to comply with treatment and follow-up schedule
* Women who may be pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | Short-term outcome 1 week
  Neck Disability Index (NDI) is a disease-specific outcome measure specifically used in patients with neck pain. The NDI has been shown to be reliable and valid in individuals with mechanical neck pain.

SECONDARY OUTCOMES:
Global Rating of Change (GROC) | Short-term outcome 1 week
  The Global Rating of Change is a outcome measure used to assess patient perceived recovery following interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Masaracchio, PT, DPT, PhD(c), OCS, SCS, Principal Investigator — Masefield Cavallaro Therapy
Locations (2):
- United States (2):
  - Long Island University, Brooklyn, New York
  - Masefield Cavallaro Physical Therapy, Brooklyn, New York